CLINICAL TRIAL: NCT04569890
Title: Study on the Treatment Strategy of Patients With Rheumatoid Arthritis During Pregnancy, a Randomized Control Trial in China
Brief Title: Treatment of Pregnancy RA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: treatment of pregnancy RA
Record Dates: First submitted 2020-09-20; First posted 2020-09-30 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis; Pregnancy Related
Keywords: Certolizumab; Hydroxychloroquine
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Hydroxychloroquine; Prednisone

STUDY DESIGN:
Intervention Model Description: Central random. Statistical experts from a third-party company not involved in the study will generate a random number table by computer system. The patients will be numbered according to their visiting order, and 1:1 allocated according to the random data table.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor and data analyst blindness. To avoid bias, physicians who assess disease activity will be blinded. Participants are required not to discuss their treatment allocation with physicians at each visit. The success of the blind method will be judged by requiring the assessors to determine the treatment allocation of participants after each visit. When the database is locked, the statistician will carry on the data analysis in the hidden of allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CZP (Experimental): Certolizumab pegol: subcutaneous CZP at 200mg twice a week.
  Interventions: Drug: Certolizumab Pegol 200 MG/ML [Cimzia]
- GC+HCQ (Active Comparator): Hydroxychloroquine: HCQ at 200mg daily, and if tolerated, escalated to 400 mg daily.
  Glucocorticoid: continuous usage GC at 10mg a day from Week 0 to Week 52.
  At 24 week, non-responders (ΔDAS28<0.6) will switch to the other group. Participants switched to CZP group will taper their dose of GC gradually, if they have an improvement in disease activity (two successive DAS28<2.6). If participants have a disease flare (increased DAS28>0.6) during a reduction in corticosteroid dose, then they will resume their previous dose. Weekly step-down GC scheme: 10mg-7.5mg-5mg-2.5mg-0mg.
  Interventions: Drug: Hydroxychloroquine; Drug: Prednisone

INTERVENTIONS:
Drug: Certolizumab Pegol 200 MG/ML [Cimzia] — CZP 200mg twice a week subcutaneous.
  Arms: CZP
Drug: Hydroxychloroquine — 400mg HCQ orally daily
  Arms: GC+HCQ
Drug: Prednisone — 10mg GC orally daily
  Arms: GC+HCQ

SUMMARY:
It is important to control the disease of pregnant women with rheumatoid arthritis to ensure the fetal and maternal health. Frequent disease flare can increase the risk of adverse pregnancy outcomes, including abortion, premature delivery and low birth weight. However, there is no scientific and standardized treatment strategy for RA during pregnancy. About 50% of RA patients need treatment during pregnancy. Tumor necrosis inhibitor (TNFi) is an effective treatment, which can significantly improve the symptoms of RA during pregnancy. However, in order to avoid placental metastasis, TNFi is usually stopped in early pregnancy. Certolizumab pegol (CZP) is a PEGylated, Fc-free TNFi, which does not bind FcRn and is consequently not expected to undergo FcRn-mediated transfer across the placenta. Therefore, it can not transfer through placenta into FcRn and is approved to treat RA during pregnancy. This study focuses on patients with RA who consider pregnancy. We compared the efficacy, safety and economy of CZP and glucocorticoids combined with hydroxychloroquine by a randomized controlled trial.

DETAILED DESCRIPTION:
In this study, a randomized controlled study was conducted to compare the efficacy, safety and economy of CZP and glucocorticoids combined with hydroxychloroquine in the treatment of RA patients who consider pregnancy. Informed consent must be obtained for the patients to be screened.

Random method: central random.

Blinding method: assessor and data analyst blindness.

Follow-up: every 4 week.

First endpoint: 24 week.

Second endpoint: 52 week.

Safety endpoint: 24 weeks postpartum.

Missing data: core data related to treatment and disease activity are not allowed to be missing, and other data are supplemented by the last observation value.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of RA, as defined by 2010 ACR/EULAR criteria
2. DAS 28∙ESR<2.6 under the treatment of DMARDs
3. Subjects consider pregnancy, but not pregnant yet
4. Participant expects to continue CZP therapy throughout pregnancy and for at least 24 weeks postpartum
5. Participant has a negative interferon gamma release assay (IGRA) or tuberculin skin test (TST) within the prior 6 months, and there has been no change in the study participant's clinical status, or social, family, or travel history. Participants with documented Bacillus Calmette-Guérin (BCG) vaccine and at low risk for tuberculosis (TB) may enroll without having a TB test performed

Exclusion Criteria:

1. Participant has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the study participant's ability to participate in this study
2. Participant is not permitted to enroll into the study if she meets any of the following TB exclusion criteria:(1) Known active TB disease; (2) History of active TB involving any organ system; (3) Latent TB infection; (4) High risk of acquiring TB infection; (5) Current nontuberculous mycobacterial (NTM) infection or history of NTM infection (unless proven to be fully recovered)
3. Study participant is taking a prohibited medication or has taken a prohibited medication
4. Live vaccine(s) within 1 month prior to Screening, or plans to receive such vaccines during the study
5. Study participant has any clinically significant pregnancy-related clinical or test abnormality, as judged by the investigator
6. Study participant had a positive or indeterminate interferon gamma release assay (IGRA) or tuberculin skin test (TST) at Screening. In case of indeterminate result, a retest is allowed if time permits; 2 results of indeterminate require exclusion of the study participant

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease Activity | 24 week
  Proportion of DAS28 remission. In principle, the score of das28-esr should be used. If there is data missing, das28-crp can be used. All patients have either complete das28-esr data or complete das28-crp data.

SECONDARY OUTCOMES:
ACR20 | 52 week
  Proportion of ACR20 improvement.
ACR50 | 52 week
  Proportion of ACR50 improvement.
ACR70 | 52 week
  Proportion of ACR70 improvement.
Time to remission | 52 week
MHAQ | 52 week
  The Modified Health Assessment Questionnaire (MHAQ), reduced the number of items from 20 in the original HAQ to eight, and improved the feasibility in clinical practice when screening patients. The MHAQ score is calculated as the mean of the scores for each activity. Total score is between 0.0-3.0, in 0.125 increments. Higher scores indicate worse function and greater disability. MHAQ scores <0.3 are considered normal.
EQ-5D | 52 week
  Health quality assessed by EuroQol five dimensions questionnaire. It is a preference-based measure that can be regarded as a continuous outcome scored on a -0.59 to 1.00 scale, with 1.00 indicating 'full health' and 0 representing dead.
Time to pregnancy | 52 week
Pregnancy rate | 52 week
Pregnancy outcomes | 0-52 week
  Pregnancy will end with live birth, stillbirth, spontaneous abortion or therapeutic abortion.

CONTACTS AND LOCATIONS:
Overall Officials: Liangjing Lu, doctor, Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Email the researchers for details.

REFERENCES:
- [Result] Mariette X, Forger F, Abraham B, Flynn AD, Molto A, Flipo RM, van Tubergen A, Shaughnessy L, Simpson J, Teil M, Helmer E, Wang M, Chakravarty EF. Lack of placental transfer of certolizumab pegol during pregnancy: results from CRIB, a prospective, postmarketing, pharmacokinetic study. Ann Rheum Dis. 2018 Feb;77(2):228-233. doi: 10.1136/annrheumdis-2017-212196. Epub 2017 Oct 13. PMID 29030361
- [Result] Forger F, Zbinden A, Villiger PM. Certolizumab treatment during late pregnancy in patients with rheumatic diseases: Low drug levels in cord blood but possible risk for maternal infections. A case series of 13 patients. Joint Bone Spine. 2016 May;83(3):341-3. doi: 10.1016/j.jbspin.2015.07.004. Epub 2015 Nov 23. PMID 26617214
- [Result] Clowse MEB, Scheuerle AE, Chambers C, Afzali A, Kimball AB, Cush JJ, Cooney M, Shaughnessy L, Vanderkelen M, Forger F. Pregnancy Outcomes After Exposure to Certolizumab Pegol: Updated Results From a Pharmacovigilance Safety Database. Arthritis Rheumatol. 2018 Sep;70(9):1399-1407. doi: 10.1002/art.40508. Epub 2018 Jul 22. PMID 29623679